CLINICAL TRIAL: NCT05307718
Title: Pharmacogenomics in Prediction of Cardiovascular Drugs Adverse Reaction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinical Hospital Centre Zagreb (Other)
Collaborators: University of Zagreb School of Medicine (Unknown); Croatian Science Foundation (Other Government)
Responsible Party: Principal Investigator, Livija Šimičević, Livija Simicevic, Clinical Hospital Centre Zagreb
Other Study IDs: UIP-2020-02-8189
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Pharmacogenetics; Drug-Related Side Effects and Adverse Reactions; Cardiovascular Drugs
Keywords: Pharmacogenetics; adverse drug reactions; statins; DOAK; platelet aggregation inhibitors
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Factor Xa Inhibitors; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The basic cohort: The subjects with the newly indicated indication for use: NOAC; platelet aggregation inhibitors from the P2Y12 receptor antagonist group; and HMG-CoA reductase inhibitors (statins
  Interventions: Drug: Oral Anticoagulant, Direct-Acting
- Cases: Cases will be subjects who have observed ADRs during follow-up: bleeding that meets the criteria of "major" or "non-major, clinically relevant bleeding (for anticoagulants and platelet aggregation inhibitors); muscle or liver lesions (for statins); any other serious ADR.
  Interventions: Drug: Oral Anticoagulant, Direct-Acting
- Controls: Controls will be subjects in whom no ADRs were observed during the study
  Interventions: Drug: Oral Anticoagulant, Direct-Acting

INTERVENTIONS:
Drug: Oral Anticoagulant, Direct-Acting — Newly indicated indication for use: DOAC; platelet aggregation inhibitors from the P2Y12 receptor antagonist group; and HMG-CoA reductase inhibitors (statins); as monotherapy or without restriction with respect to any other concomitant pharmacotherapy. Subjects will be followed up during regular visits.
  Other Names: HMG-CoA reductase inhibitors; platelet aggregation inhibitors from the P2Y12 receptor antagonist group

SUMMARY:
The research is planned as a prospective nested case-control study. The plan is to recruit about 1,200 consecutive subjects whose pharmacotherapy involves the drug(s) of interest within 4.5 years. The basic cohort - the subjects with the newly indicated indication for use: NOAC; platelet aggregation inhibitors from the P2Y12 receptor antagonist group; and HMG-CoA reductase inhibitors (statins); as monotherapy or without restriction with respect to any other concomitant pharmacotherapy. The ADRs will be analysed by CR by: age, gender, expectancy, severity, association, type (mechanism of event), and outcome, according to the classification of organ systems as well as association with the phenotype. Criteria for bleeding associated with the use of anticoagulant and antiplatelet therapy have been defined; as well as the myotoxicity and hepatotoxicity associated with statin therapy. Samples will be tested for biochemical, haematological, coagulation standard parameters and pharmacogenetic analyses of relevant genes depending on the used therapy. Pharmacogenetic analysis will be performed to genotype the polymorphisms of relevant pharmacogenes: Biological samples and clinical data will be anonymized plus all records of ADRs and other clinical variables will be protected. Possible drug-drug and drug-drug-gene interactions will be evaluated using the Clinical Decision Support System (CDSS) of Lexicomp, PharmGKB, the Flockhart Table, and other systems including panel consensus methods to determine the likelihood of an ADR being associated with drug interactions, and determine whether drug interactions contributed to the occurrence of ADRs to administered CV pharmacotherapy in subjects with variant pharmacogenes of interest (drug-drug-gene interaction). The overall project objective is to determine which pharmacogenes variants, together with clinical parameters, can be used as predictors of CV drug ADRs and are good candidates for inclusion in the clinical diagnostic panel for pre-emptive PGx testing.

ELIGIBILITY:
Inclusion Criteria:

a) age 18 years or older; b) a new indication for the administration of any of the medicinal products of primary interest (NOAC, clopidogrel, prasugrel, ticagrelor, statins) for which at least a 3-month administration is predicted; c) signed informed consent (for repeated evaluations and donation of blood samples for genetic and eventual pharmacokinetic analysis).

Exclusion Criteria:

the existence of contraindications to the medicines of primary interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The primary cohort is represented by subjects who have a new indication for the administration of a) new oral anticoagulants (NOAC); b) platelet aggregation inhibitors from the P2Y12 receptor antagonist group (clopidogrel, prasugrel, ticagrelor); c) an HMG-CoA reductase inhibitor (statins); for the purpose of treatment or prophylaxis for at least 3 months; as monotherapy or without restriction with respect to any other concomitant pharmacological therapy.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2025-12-14 (Estimated); Study Completion 2025-12-14 (Estimated)

PRIMARY OUTCOMES:
The overall project objective is to determine which pharmacogenes variants, together with clinical parameters, can be used as predictors of CV drug ADRs | 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Bozina, PhD, Principal Investigator — University of Zagreb, Schooll of Medicine
Locations (1):
- UHC Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bozina T, Ganoci L, Simicevic L, Vrkic Kirhmajer M, Mucalo I, Samardzic J, Palic J, Sliskovic AM, Trkulja V. Pharmacogenomics in the prediction of adverse effects of cardiovascular drugs: the PGx-CardioDrug project. Croat Med J. 2026 Jan 5;66(6):446-455. doi: 10.3325/cmj.2025.66.446. PMID 41520206
- See also: Project web site — https://mef.unizg.hr/znanost/istrazivanje/web-stranice-projekata/projekt-hrzz-pgx-cardiodrug/